CLINICAL TRIAL: NCT03765905
Title: Evaluation of Serum Scube-1 Scube-2 and Scube-3 Levels in Patients With Polikistik Over Syndrome ,
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Suleyman Guven, Clinical professor, Karadeniz Technical University
Other Study IDs: Karadeniz Technical University
Record Dates: First submitted 2018-06-22; First posted 2018-12-05 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; SCUBE; Cardiovascular disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS diagnosis area: The study group consisted of 40 reproductive age women between 18th and 35th years old women who were PCOS diagnosis (according to the 2003 Rotherdam criteria)
  Interventions: Diagnostic Test: study
- PCOS is not diagnosed: Forty patients who did not have any complaints between the ages of 18-35 who applied to the gynecology policlinic as a control group but who had no PCOS orany other systemic problems and were similar in terms of age group and body mass index were included in the study after being approved for participation in the study
  Interventions: Diagnostic Test: study

INTERVENTIONS:
Diagnostic Test: study — Scube-1 scube-2 scube-3

SUMMARY:
The aim of this study is to investigate serum SCUBE-1 and SCUBE-3 levels in PCOS and non-PCOS cases compared with non-PCOS healthy controls with similar age and body mass index

DETAILED DESCRIPTION:
The aim of this study was to investigate serum SCUBE1 and SCUBE3 levels in PCOS and non-PCOS cases compared with non-PCOS healthy controls with similar age and body mass index.

This will be a prospective clinical laboratory study,It will include women with PCOS diagnosis (according to the 2003 Rotherdam criteria). 40 cases of reproductive age will be included in the study group, which will be included in the survey after being approved for participation in the survey from field trials. Forty patients who will not have any complaints between the ages of 18-35 who will apply to the gynecology policlinic as a control group but who had no PCOS o rany other systemic problems and will be similar in terms of age group and body mass index will be included in the study after being approved for participation in the study. From the study and control group, 5 mL of blood will be taken from the untreated biochemical tube for serum SCUBE1 SCUBE2 SCUBE3. The blood samples will be centrifuged at 1000 g for 10 minutes and the serum fraction will be obtained and the serum will be stored at -80 ° C to be stored until the day of the tube operation. Serum SCUBE1, SCUBE2 SCUBE3 levels will be measured using ELISA kits. ,

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of PCOS
* 18-35 years old

Exclusion Criteria

* Endocrinopathies (including diabetes mellitus, hyperprolactinemia, Cushing's disease and congenital adrenal hyperplasia), systemic disease (eg asthma), collagen disorder, hypercholesterolemia, sickle cell anemia or neoplasm,
* Coronary artery disease , angina or myocardial infarction, or any known vascular, infectious, or inflammatory disease, including hypertension, coronary arterioscitis, and electrocardiographic changes;
* Use of any medication (e.g., insulin sensitizing drugs, oral contraceptives, antiandrogens, statins, aspirin, corticosteroids and gonadotropin releasing hormone agonists and antagonists) within the previous 3 months;
* Abnormal serum albumin concentration (normal concentration, 30-55 g / l),
* Abnormal troponin I concentration,
* Present smoker,
* Abnormal renal, hepatic and thyroid function test results;
* Refusing to participate in the work.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 women diagnosed with PCOS between the ages of 18-35
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Serum SCUBE 1 | 01.01.2017-31.12.2017
  Serum scube1 in microgram
Serum SCUBE 2 | 01.01.2017-31.12.2017
  Serum scube2 in microgram
Serum SCUBE 3 | 01.01.2017-31.12.2017
  Serum scube3 in microgram

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Güven, Prof, Principal Investigator — Karadeniz TU Medicine Faculty
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided